CLINICAL TRIAL: NCT06877299
Title: Low-Dose Radiation + Stereotactic Body Radiotherapy Followed by Tislelizumab Plus Platinum-based Chemotherapy As Neoadjuvant Therapy in Patients With Resectable StageⅡA-ⅢB Non-small Cell Lung Cancer
Brief Title: Low-Dose Radiation + SBRT + Tislelizumab Plus Platinum-based Chemotherapy in Stage ⅡA-ⅢB Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, You Lu, Chair of Division of Thoracic Tumor Multimodality Treatment, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IHC-003
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer; Non-small Cell Lung Cancer
Keywords: Neoadjuvant; Low Dose Radiotherapy; Stereotactic Body Radiotherapy; Immunotherapy; NSCLC
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery; tislelizumab; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiation therapy combined with PD-1 inhibitor and chemotherapy group (Experimental): Low-Dose Radiation(2Gy*2-3d) +Stereotactic body radiation therapy (10Gy*3d) followed by Tislelizumab (200mg) with platinum-based doublet chemotherapy administered pre-operatively every 3 weeks for 3 cycles before surgical resection.
  Interventions: Drug: Low-Dose Radiation(LDRT) + Stereotactic body radiotherapy (SBRT)

INTERVENTIONS:
Drug: Low-Dose Radiation(LDRT) + Stereotactic body radiotherapy (SBRT) — Low-Dose Radiation(LDRT) + Stereotactic body radiotherapy (SBRT)
  Other Names: Drug: Tislelizumab; Drug: Chemotherapy

SUMMARY:
This phase II study aims to evaluate the efficacy and safety of low-dose radiation + SBRT + Tislelizumab plus platinum-based chemotherapy as neoadjuvant therapy for stage II-III non-small cell lung cancer.

DETAILED DESCRIPTION:
All eligible patients will receive LDRT combined with partial SBRT, followed by PD-1 inhibitors plus platinum-based chemotherapy, initiated within 7 days after completing radiation. PD-1 inhibitors and chemotherapy will be administered at the recommended doses according to the instruction manual every 3 weeks, with 3 cycles planned as neoadjuvant therapy. Surgery will be performed within 4 to 6 weeks (+7 days) after completing the final cycle of immunochemotherapy.

Main objective and endpoint: the rate of pathological complete response (pCR) in the resected primary tumor and lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75 years;
2. Patients with untreated stage IIA-IIIB non-small cell lung cancer, diagnosed cytologically or histologically (according to the AJCC 9th edition of thoracic tumor staging);
3. Pulmonary lesions will be assessed as resectable or potentially resectable by a multidisciplinary team, including a thoracic surgeon;
4. At least one imaging-measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1);
5. Ability to provide tumor tissue or cell wax blocks that meet quality control standards for PD-L1 expression testing.

Exclusion Criteria:

1. The pathology is small cell lung cancer (SCLC), including lung cancer mixed with SCLC and non-small cell lung cancer (NSCLC)；
2. Patients with known EGFR-sensitive mutations or ALK fusion.
3. Previously received the following therapies: anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or another drug that stimulates or synergistically inhibits T cell receptors;
4. Subjects with any known or suspected autoimmune disorder or immunodeficiency, with the following exceptions: hypothyroidism, hormone therapy is not needed, or well controlled at physiological dose; controlled type I diabetes;
5. Active infection requiring systemic treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-04 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
pCR rate | From date of enrollment until one month after resection
  pCR is defined as the absence of residual invasive cancer on hematoxylin and eosin stained slides of the resected lung specimen and lymph nodes following completion of neoadjuvant therapy

SECONDARY OUTCOMES:
MPR rate | From date of enrollment until one month after resection
  mPR is defined as ≤10% viable tumor cells in the resected primary tumor and all resected lymph nodes.
R0-resection rate | From date of enrollment until one month after resection
Event-free survival (EFS) | up to 2 years
  EFS is defined as the time from enrollment to radiographic disease progression, local progression precluding surgery, inability to resect the tumor, local or distant recurrence, or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: You Lu, MD. PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- West China Hospital of Sichuan University, Chengdu, China, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao ZR, Liu SL, Zhou T, Chen G, Long H, Su XD, Zhang X, Fu JH, Lin P, Zhang LJ, Rong TH, Wu JD, Li ZC, Su HL, Chen JY, Yang YP, Lin YB, Xi M, Yang H. Stereotactic body radiotherapy with sequential tislelizumab and chemotherapy as neoadjuvant therapy in patients with resectable non-small-cell lung cancer in China (SACTION01): a single-arm, single-centre, phase 2 trial. Lancet Respir Med. 2024 Dec;12(12):988-996. doi: 10.1016/S2213-2600(24)00215-7. Epub 2024 Sep 18. PMID 39305910
- [Background] Yue D, Wang W, Liu H, Chen Q, Chen C, Liu L, Zhang P, Zhao G, Yang F, Han G, Cheng Y, Yu B, Yang Y, Chen H, Jiang J, Tan L, Xu S, Mao N, Hu J, Zhang L, Yao B, Wang S, Wang RH, Zheng W, Wang C; RATIONALE-315 investigators. Perioperative tislelizumab plus neoadjuvant chemotherapy for patients with resectable non-small-cell lung cancer (RATIONALE-315): an interim analysis of a randomised clinical trial. Lancet Respir Med. 2025 Feb;13(2):119-129. doi: 10.1016/S2213-2600(24)00269-8. Epub 2024 Nov 21. PMID 39581197
- [Background] Forde PM, Spicer J, Lu S, Provencio M, Mitsudomi T, Awad MM, Felip E, Broderick SR, Brahmer JR, Swanson SJ, Kerr K, Wang C, Ciuleanu TE, Saylors GB, Tanaka F, Ito H, Chen KN, Liberman M, Vokes EE, Taube JM, Dorange C, Cai J, Fiore J, Jarkowski A, Balli D, Sausen M, Pandya D, Calvet CY, Girard N; CheckMate 816 Investigators. Neoadjuvant Nivolumab plus Chemotherapy in Resectable Lung Cancer. N Engl J Med. 2022 May 26;386(21):1973-1985. doi: 10.1056/NEJMoa2202170. Epub 2022 Apr 11. PMID 35403841
- [Result] Zhou X, Zhou L, Yao Z, Huang M, Gong Y, Zou B, Zhu J, Liu Y, Peng F, Zhang Y, Yu M, Li Y, Na F, Wu Y, Kang K, Xiu W, Zhang X, Zhou L, Xu Y, Wang J, Wang Y, Yang X, Wu Y, Li R, Zhang Y, Yang Z, Zhou Z, Bai J, Yi X, Tong R, Yin L, Chen C, Niedermann G, Lu Y, Xue J. Safety and Tolerability of Low-Dose Radiation and Stereotactic Body Radiotherapy + Sintilimab for Treatment-Naive Stage IV PD-L1+ Non-Small Cell Lung Cancer Patients. Clin Cancer Res. 2023 Oct 13;29(20):4098-4108. doi: 10.1158/1078-0432.CCR-23-0315. PMID 37581611
- [Result] Yin L, Xue J, Li R, Zhou L, Deng L, Chen L, Zhang Y, Li Y, Zhang X, Xiu W, Tong R, Gong Y, Huang M, Xu Y, Zhu J, Yu M, Li M, Lan J, Wang J, Mo X, Wei Y, Niedermann G, Lu Y. Effect of Low-Dose Radiation Therapy on Abscopal Responses to Hypofractionated Radiation Therapy and Anti-PD1 in Mice and Patients With Non-Small Cell Lung Cancer. Int J Radiat Oncol Biol Phys. 2020 Sep 1;108(1):212-224. doi: 10.1016/j.ijrobp.2020.05.002. Epub 2020 May 15. PMID 32417411